CLINICAL TRIAL: NCT05754164
Title: Attention Control Training for the Prevention of PTSD in Firefighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Collaborators: Kungming Training Corps of National Fire and Rescue Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XF002
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: PTSD
Keywords: PTSD; Attention Control Training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control Training (Experimental): The Dot-Probe Paradigm was utilized within the Attention Bias Modification procedure. The training sessions were comprised of 80 trials, which included facial expression photos depicting happiness, neutrality, and sadness, sourced from four male and four female actors. A fixed cross (+) was presented on the computer screen's center for a duration of 500 milliseconds before each stimulus display, followed by the presentation of two images portraying distinct emotional expressions, which persisted for 500 milliseconds. After the disappearance of the images, an arrow appeared in the location where they had been displayed, and participants were instructed to select the arrow that corresponded with the presented arrow. In the ABM procedure, the arrow was consistently presented following the display of a more positive facial expression, such that in the instance of a sad-neutral face pair, the arrow would always appear in the location of the neutral facial expression image.
  Interventions: Behavioral: Attention Control Training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Attention Control Training — Mobile app-based attention control training is an effective training method that can help people improve their ability to control attention. It is generally recommended to undergo 4 weeks of training, with 3-4 sessions per week and one day between each session. The specific operational method of this training may vary depending on different applications, but generally, training is presented in the form of a series of tasks. These tasks may involve aspects such as focusing attention, inhibiting interference, and reacting quickly.
  Arms: Attention Control Training

SUMMARY:
The study aimed to examine the effect of Attention Control Training (ACT) intervention on reducing PTSD symptoms in firefighters. The study was a randomized controlled trial carried out in Kunming, China, and involved the recruitment of 180 active firefighters as participants. The intervention lasted for an 8-week duration, during which participants participated in ACT exercises delivered through a smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* being an active firefighter and aged between 18 and 50
* with no history of severe PTSD

Exclusion Criteria:

* having suicidal ideation or intent
* having an active psychotic disorder other than PTSD
* prior participation in a cognitive-behavioral intervention
* concurrent participation in another study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist-Civilian Version | Baseline
  The PCL-C scale (Posttraumatic Stress Disorder Checklist-Civilian Version) is a self-report questionnaire that assesses symptoms of post-traumatic stress disorder (PTSD) in adults who have experienced a traumatic event. The PCL-C is based on the DSM-IV criteria for PTSD and includes 17 items that correspond to the three symptom clusters of PTSD: re-experiencing, avoidance/numbing, and hyperarousal.
  The PCL-C scale is widely used in both clinical and research settings to screen for and assess PTSD symptoms. It is a quick and easy-to-administer tool that can help healthcare professionals identify individuals who may need further evaluation and treatment for PTSD. The PCL-C can also be used to monitor the severity of PTSD symptoms over time and to evaluate the effectiveness of PTSD treatments.
Posttraumatic Stress Disorder Checklist-Civilian Version | Immediately Post-intervention
  The PCL-C scale (Posttraumatic Stress Disorder Checklist-Civilian Version) is a self-report questionnaire that assesses symptoms of post-traumatic stress disorder (PTSD) in adults who have experienced a traumatic event. The PCL-C is based on the DSM-IV criteria for PTSD and includes 17 items that correspond to the three symptom clusters of PTSD: re-experiencing, avoidance/numbing, and hyperarousal.
  The PCL-C scale is widely used in both clinical and research settings to screen for and assess PTSD symptoms. It is a quick and easy-to-administer tool that can help healthcare professionals identify individuals who may need further evaluation and treatment for PTSD. The PCL-C can also be used to monitor the severity of PTSD symptoms over time and to evaluate the effectiveness of PTSD treatments.
Patient Health Questionnaire-9 | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) was utilized to assess symptoms of depression. The PHQ-9 is a selfreport questionnaire comprising 9 items, with a score range of 0-27, measuring depression-related symptoms experienced in the past two weeks
Patient Health Questionnaire-9 | Immediately Post-intervention
  The Patient Health Questionnaire-9 (PHQ-9) was utilized to assess symptoms of depression. The PHQ-9 is a selfreport questionnaire comprising 9 items, with a score range of 0-27, measuring depression-related symptoms experienced in the past two weeks
Generalized Anxiety Disorder 7-item scale | Baseline
  The GAD-7 scale (Generalized Anxiety Disorder 7-item scale) is a self-report questionnaire used to assess symptoms of generalized anxiety disorder (GAD) in adults. The GAD-7 includes seven items that correspond to the DSM-IV criteria for GAD, such as feeling nervous, anxious or on edge, worrying too much, and having trouble relaxing.
  The GAD-7 is a brief and easy-to-use tool that has been validated in various settings, including primary care, psychiatric clinics, and community-based samples. It is designed to help healthcare professionals screen for and assess the severity of GAD symptoms in their patients.
Generalized Anxiety Disorder 7-item scale | Immediately Post-intervention
  The GAD-7 scale (Generalized Anxiety Disorder 7-item scale) is a self-report questionnaire used to assess symptoms of generalized anxiety disorder (GAD) in adults. The GAD-7 includes seven items that correspond to the DSM-IV criteria for GAD, such as feeling nervous, anxious or on edge, worrying too much, and having trouble relaxing.
  The GAD-7 is a brief and easy-to-use tool that has been validated in various settings, including primary care, psychiatric clinics, and community-based samples. It is designed to help healthcare professionals screen for and assess the severity of GAD symptoms in their patients.
Attention Bias Score | Baseline
  To quantify attention bias, response times (RTs) were analyzed in accordance with the established procedure to calculate the attention bias score (ABS). Trials characterized by inaccurate responses or RTs of exceptional brevity (<150ms) or prolonged duration (>1200ms) were disregarded. The computation of attention bias entailed determining the discrepancy between the mean RT in response to relatively positive stimuli and the mean RT in response to relatively negative stimuli. A preference for happy faces was indicated by an average RT for happy facial expressions that were shorter than the average RT for neutral or sad facial expressions.
Attention Bias Score | Immediately Post-Intervention
  To quantify attention bias, response times (RTs) were analyzed in accordance with the established procedure to calculate the attention bias score (ABS). Trials characterized by inaccurate responses or RTs of exceptional brevity (<150ms) or prolonged duration (>1200ms) were disregarded. The computation of attention bias entailed determining the discrepancy between the mean RT in response to relatively positive stimuli and the mean RT in response to relatively negative stimuli. A preference for happy faces was indicated by an average RT for happy facial expressions that were shorter than the average RT for neutral or sad facial expressions.
Attention Bias Variability | Baseline
  To quantify attention-bias variability (ABV), the experimental data were divided into 8 segments, and attention-bias scores were computed for each segment. Subsequently, the standard deviation of attention-bias scores across segments was determined, and this value was divided by all trials ABS to account for ABS variability.
Attention Bias Variability | Immediately Post-Intervention
  To quantify attention-bias variability (ABV), the experimental data were divided into 8 segments, and attention-bias scores were computed for each segment. Subsequently, the standard deviation of attention-bias scores across segments was determined, and this value was divided by all trials ABS to account for ABS variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Training Corps of the National Fire and Rescue Administration, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No